CLINICAL TRIAL: NCT06023758
Title: A Multicenter II Study to Compare KN026 and KN046 Versus Oxaliplatin, Capecitabine Combined KN026 and KN046 in Patients With HER2-positive Locally Advanced Resectable Gastric Cancer or Gastroesophageal Junction Adenocarcinoma.
Brief Title: Phase 2 Trial of KN026+KN046±XELOX in HER2-positive Locally Advanced GC
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Peking University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: KHER2-001
Record Dates: First submitted 2023-08-08; First posted 2023-09-05 (Actual); Last update posted 2024-05-10 (Actual); Status verified 2023-08

CONDITIONS: HER2-positive Locally Advanced Resectable Gastric Cancer
MeSH Terms: interventions — XELOX

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- KN026 combined with KN046 (Experimental): KN026 combined with KN046
  Interventions: Drug: KN026; Drug: KN046
- KN026，KN046 and XELOX (Experimental): KN026，KN046 and XELOX
  Interventions: Drug: KN026; Drug: KN046; Drug: XELOX

INTERVENTIONS:
Drug: KN026 — KN026：30 mg/kg Q3W
Drug: KN046 — KN046：5 mg/kg Q3W
Drug: XELOX — Oxaliplatin 130mg/m2 d1，Capecitabine 1000mg/m2 d1-14，Q3W
  Arms: KN026，KN046 and XELOX

SUMMARY:
This is a multicenter II study to compare KN026 and KN046 versus Oxaliplatin, Capecitabine combined KN026 and KN046 in patients with HER2-positive locally advanced resectable gastric cancer or gastroesophageal junction adenocarcinoma.

DETAILED DESCRIPTION:
KN026 is an anti-HER2 bispecific antibody that can simultaneously bind two non-overlapping epitopes of HER2, resulting in dual HER2 signaling blockade.KN046 is a PD-L1 - CTLA-4 bispecific antibody. The trial consists of two groups. All subjects will be treated with KN026 at 30 mg/kg Q3W in combination with KN046 at 5 mg/kg Q3W in Group 1. If the statistical hypothesis is not met in Group 1, patients will be enrolled in Group 2. Patients in group 2 will receive KN026+KN046+XELOX.

ELIGIBILITY:
Inclusion Criteria:

* The subject can understand the informed consent, voluntarily participate and sign the informed consent ;
* Subjects are older than or equal to 18 years old and younger than or equal to 75 years old on the day of signing the informed consent；
* Histologically or cytologically confirmed, locally advanced HER2-positive gastric cancer or gastroesophageal junction adenocarcinoma.
* ECOG score 0 or 1;
* Left ventricular ejection fraction (LVEF) ≥ 50% at baseline as determined by either ECHO (preferred) or MUGA;
* Liver function met the following criteria within 7 days prior to initial administration:

Total bilirubin ≤1.0x ULN (Gilbert's syndrome, or total bilirubin ≤1.5x ULN in liver metastases); Aminotransferase (ALT/AST) ≤1.5x ULN (liver metastatic subjects ≤3xULN); -Renal function within 7 days prior to initial administration: serum creatinine ≤1.5x ULN and serum creatinine clearance ≥60mL/min (according to Cockcroft-Gault Formula calculation);

* Bone marrow function met the following criteria within 7 days prior to initial administration: Hemoglobin ≥90 g/L; Neutrophil absolute count ≥1.5 x 109/L; Platelet count ≥100x 109/L; INR or PT≤1.5x ULN, and aPTT≤ 1.5x ULN;
* Life expectancy >3 months;
* The subjects are able and willing to follow the visits, treatment plans, laboratory tests, and other study-related procedures specified in the study protocol

Exclusion Criteria:

* Existence of other active malignant tumors within 5 years or at the same time. Plan to perform or have undergone an organ or bone marrow transplant. Myocardial infarction and poorly controlled arrhythmias occurred within 6 months prior to the first dose.
* Existence of grade III - IV cardiac disorders defined by the NYHA or echocardiogram shows: LVEF (left ventricular ejection fraction) < 50%.
* Human immunodeficiency virus (HIV) infection.
* Patients with active tuberculosis.
* Patient with previous or current interstitial pneumonia, pneumoconiosis, radiation pneumonitis, drug-associated pneumonia, severely impaired lung function, etc.
* Patients who have previously received other antibody/drug treatments for immune checkpoints, such as PD-1, PD-L1, and CTLA4 treatments.
* Have diseases that may increase the risk of participating in the study and using the study medications, or other severe, acute, and chronic diseases and therefore are judged by the investigator to be unsuitable for clinical studies.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2023-09-22 (Actual); Primary Completion 2025-09-01 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
pCR rate | up to 2 years
  Pathological complete response (pCR) rate (assessed by central pathology laboratory and the site)

SECONDARY OUTCOMES:
Event-free survival (EFS) | from enrollment until firstly confirmed and recorded disease progression or death，assessed up to 3 years
  Event-free survival (assessed by the investigator per RECIST v1.1 criteria)
Disease-free survival (DFS) | from the start of surgery to disease recurrence or death (for any reason)，assessed up to 3 years
  Disease-free survival (assessed by the investigator per RECIST v1.1 criteria)
overall survival (OS) | From date of randomization until the date of death from any cause, assessed up to 5 years
  overall survival

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Cancer Hospital, Beijing, Beijing Municipality, China